CLINICAL TRIAL: NCT02700412
Title: University of Alabama at Birmingham (UAB) Adult CBD Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jerzy P Szaflarski, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-140826007
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2019-05

CONDITIONS: Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epidiolex 100 milligram/milliliter (mg/mL) oral solution (Experimental): Participants will receive a CBD starting dose of 5 mg/kg/day in twice daily dosing and titrate by 5 mg/kg/2 weeks up to 25 mg/kg/day. Additional increases in dosing, by 5 mg/kg/day up to a maximum of 50 mg/kg/day, may be instituted at the discretion of the treating Principle Investigator (PI).
  If a subject experiences a "clinically significant" or "dose limiting" adverse event (AE) or severe adverse event (SAE) attributable to CBD, the investigator will determine if a dose reduction or taper is necessary (decreases will occur in 5 mg/kg/2 week increments or at a rate felt appropriate by the treating PI).
  Interventions: Drug: Epidiolex

INTERVENTIONS:
Drug: Epidiolex — Epidiolex oral solution (100 mg/mL CBD concentration) with inactive ingredients including anhydrous ethanol, sesame seed oil, strawberry flavor, and sucralose).
  Other Names: Cannabidiol; CBD

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Epidiolex at various doses between 5 mg/kg/day and 50 mg/kg/day as an additional (add-on) drug for treating debilitating, drug-resistant epilepsy.

DETAILED DESCRIPTION:
The specific goals of this phase 1 dose finding study, conducted in consecutively enrolled patients 18 years of age and older, are to prospectively and longitudinally assess the safety and tolerability, including cognitive effects, of Cannabidiol (CBD) at various doses between 5 mg/kg/day and 25 mg/kg/day, with additional titration in some cases up to 50 mg/kg/day. In order to participate in the study, participants will need to fulfill the inclusion and exclusion criteria.

The goal of the study is to fulfill the mandate of "Carly's Law" and to provide patients with debilitating epileptic conditions with access to CBD as an add-on treatment. Other care including routine neurological care unrelated to participation in the CBD study will need to be provided by patients' primary/current treating neurologist.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with disabling epilepsy with diagnosis confirmed by video/EEG monitoring, and
* Patient should have history of a trial of at least four anti-epileptic drugs (AEDs) including one trial of a combination of two concomitant AEDs, without successful seizure control. Vagus nerve stimulation (VNS), Responsive Neurostimulation (RNS) deep brain stimulation, or the ketogenic diet can be considered an equivalent to a drug trial,
* Between 1-4 baseline anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to submitting records for review by the CBD Treatment Approval Committee.
* VNS or RNS must be on stable settings for a minimum of 3 months,
* If on ketogenic diet, must be on stable ratio for a minimum of 3 months.
* The referring provider needs to make available for review all of the following:

  * Most recent Brain MRI report,
  * Most recent ECG report,
  * Video/EEG monitoring report confirming the diagnosis of epilepsy,
  * Evidence that the patient has failed 4 AEDs as indicated above,
  * Current Medication List
  * Patient must have at least 4 clinically countable seizures per month.
  * Seizure history to include a documented history of generalized seizures (drop attacks, atonic, tonic-clonic and/or myoclonic), focal seizures without loss of consciousness with a motor component, focal seizures with loss of consciousness, or focal seizures with secondary generalization,
  * Results of routine testing including blood work (Complete Blood Count (CBC), Comprehensive Metabolic Panel (CMP), Liver Function Tests (LFTs), renal panel, Urinary Analysis (UA), and levels of all AEDs) and digital copy of a routine EEG along with the formal written report performed within 3 months prior to submitting records for CBD Treatment Approval review. If any AED dose was adjusted within 3 months prior to submitting records for CBD Treatment Approval Committee review, level on the new dose will need to be provided. If applicable, results of any metabolic or genetic testing performed should be included in submitted records for review:
  * If applicable, documentation (including date of surgery) of prior VNS, RNS, Corpus Callosotomy, or other epilepsy surgery the patient has received.
* Age 15 years and older,
* Patients are able to keep and provide seizure calendar for at least 3 months prior to submitting records for CBD Treatment Approval Committee review. The patient will need to provide an updated calendar at the time of enrollment,
* Acceptable method of contraception (or abstinence) for women of childbearing potential and for male patients with partners of childbearing potential; female patients must have a negative urine pregnancy test on the day of initiating CBD,
* For patients who agree to participate in the optional neuroimaging sub-study, an MRI screen will be obtained to show that the patient does not have contraindication to receiving MRI/function MRI (fMRI) at 3 Tesla (e.g., metallic artifact).
* Approval for inclusion by the CBD Treatment Approval Committee.
* Current State of Alabama Resident
* Acceptable documentation of Alabama residency includes the following:

  * a state issued identification (ID), such as a driver's license, from patient or patient's parent/legally authorized representative (LAR).
  * documents showing the patient or patient's parent/LAR rents/owns property in the state,
  * state voter registration from patient or patient's parent/LAR, or
  * a recent state tax return from patient or patient's parent/LAR.

Exclusion Criteria:

* Active Psychogenic Non-Epileptic Seizures (PNES); Patients with more than 1 year freedom from PNES will not be excluded,
* Patients who are pregnant, breastfeeding, or not using acceptable methods of contraception during the course of the study and for three months thereafter,
* Male patient's partner is of child bearing potential; unless willing to ensure that they (male patients) or their partner(s) are using acceptable methods of contraception during the course of the study and for three months thereafter,
* History of substance abuse/addiction,
* Use of medical marijuana or CBD based product in the past 30 days,
* Initiation of felbamate within last 12 months,
* Allergy to CBD or any marijuana-type products,
* Alanine Aminotransferase (ALT) >5 x Upper Limit of Normal (ULN) or Aspartate Aminotransferase (AST) >5 x ULN, as seen in participant's laboratory results submitted to the CBD Treatment Approval Committee for review.
* Hemoglobin <10 or Hematocrit <30 or White Blood Count (WBC) < 2000, as seen in participant's laboratory results submitted to the CBD Treatment Approval Committee for review.
* In investigator's judgment, active medical condition/treatment that impacts study activities.
* Unable to provide consent (and no LAR),
* Unable/Failure to comply with study visits/requirements and/or instructions,
* Confirmed diagnosis for Dravet Syndrome or Lennox Gastaut Syndrome that qualifies the patient for a Greenwich (GW) Dravet Syndrome or Lennox Gastaut Syndrome randomized controlled clinical trial for which the patient is eligible pursuant to the GW clinical trial enrollment criteria unless

  * (a) there is no study that is either actively open for enrollment of patients at the University of Alabama at Birmingham (UAB) or that is expected to actively begin enrolling patients at UAB within two (2) months of the date on which the patient is screened for the UAB Pediatric CBD Program or UAB Adult CBD Program,
* Subjects with contraindications to MRI/fMRI at 3 Tesla (e.g., metallic artifact) will not be offered participation in the optional substudy.
* Primary residence in a State different than Alabama.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Szaflarski, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duncan JS, Sander JW. The Chalfont Seizure Severity Scale. J Neurol Neurosurg Psychiatry. 1991 Oct;54(10):873-6. doi: 10.1136/jnnp.54.10.873. PMID 1744641
- [Background] Pinheiro, J.C. and Bates, D.M. (2000). Mixed-Effects Models in S and S-Plus. Springer, Verlag, New York.
- [Derived] Szaflarski JP, Hernando K, Bebin EM, Gaston TE, Grayson LE, Ampah SB, Moreadith R. Higher cannabidiol plasma levels are associated with better seizure response following treatment with a pharmaceutical grade cannabidiol. Epilepsy Behav. 2019 Jun;95:131-136. doi: 10.1016/j.yebeh.2019.03.042. Epub 2019 Apr 29. PMID 31048098
- [Derived] Warren PP, Bebin EM, Nabors LB, Szaflarski JP. The use of cannabidiol for seizure management in patients with brain tumor-related epilepsy. Neurocase. 2017 Oct-Dec;23(5-6):287-291. doi: 10.1080/13554794.2017.1391294. Epub 2017 Oct 24. PMID 29063814
- See also: UAB Cannabidiol Program — http://www.uab.edu/cbd

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with treatment-resistant epilepsy in the state of Alabama were enrolled. Their primary treating neurologist provided the UAB CBD Treatment Approval Committee with the required information (found on www.uab.edu/cbd) to review. The committee either "approved/recommended" or "disapproved/not recommended" them for treatment in the study.
Pre-assignment Details: Of the total 129 participants with epilepsy ages 18 years and older screened, 80 were enrolled in this single-center, open-label study. This study was not randomized.
Groups:
- Epidiolex: The participants (or their caregivers) self-administered CBD 100mg/mL oral solution at a starting dose of 5 mg/kg/day in twice daily dosing and titrated by 5 mg/kg/2 weeks up to 25 mg/kg/day. Additional increases in dosing, by 5 mg/kg/day up to a maximum of 50 mg/kg/day, was instituted at the discretion of the treating PI.
Period: Overall Study
Arm/Group | Epidiolex
Started | 80
Completed | 47
Not Completed | 33
Not completed — Adverse Event | 6
Not completed — Death | 1
Not completed — Lack of Efficacy | 19
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for all participants who received Epidiolex at the starting dose of 5 mg/kg.
Arm/Group | Epidiolex
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8125 (13.5787)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6
  White | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Adverse Events (SAEs) (Increase in Seizure Frequency by More Than 100% Leading to Emergency Room Visit or Hospitalization).
Description: Severe adverse events (SAEs) were defined as increase in seizure frequency by more than 100% leading to emergency room visit or hospitalization. During study clinic and phone visits, adverse and severe adverse event monitoring and reporting were assessed among all participants. Data was recorded and stored in the UAB RedCap System.
Time Frame: For 1 Year following Enrollment
Population: Per protocol, after all participants have been enrolled and followed for 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidiolex
Number analyzed (Participants) | 80
Participants | 0

2. Primary Outcome: Number of Participants With Change in Resting Blood Pressure or Heart Rate by 25% if Considered Significant by Managing Neurologist.
Description: During study clinic visits, participant vital signs, including blood pressure and heart rate, were collected. Data was recorded and stored in the UAB RedCap System. Clinically significant was determined by using the Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03. Adverse events categorized as a grade 3 or above were considered clinically significant. Adverse events grade 4 or above were considered severe adverse events.
Time Frame: For 1 Year following Enrollment
Population: Per protocol, after all participants have been enrolled and followed for 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidiolex
Number analyzed (Participants) | 80
Participants
  Blood Pressure | 0
  Heart Rate | 0

3. Primary Outcome: Number of Participants With Change in Laboratory Tests Considered by Managing Neurologists as Clinically Significant.
Description: During study clinic visits, participants received laboratory testing to assess for side effects and toxicity. Data was recorded and stored in the UAB RedCap System. Laboratory testing included Complete Blood Count (CBC), Comprehensive Metabolic Panel (CMP; included Liver Function Tests (LFTs) mainly looking at alanine aminotransferase (ALT) and aspartate aminotransferase (AST)), Urine Analysis (UA), and Antiepileptic Drug (AED) levels. Clinically significant was determined by using the Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03. Adverse events categorized as a grade 3 or above were considered clinically significant. Adverse events grade 4 or above were considered severe adverse events.
Time Frame: For 1 Year following Enrollment
Population: Per protocol, after all participants have been enrolled and followed for 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidiolex
Number analyzed (Participants) | 80
Participants
  CBC: White Blood Cell (WBC) Count | 0
  CBC: Red Blood Cell (RBC) Count | 0
  CBC: Hemoglobin | 0
  CBC: Hematocrit | 0
  CBC: Platelet | 2
  CBC: Absolute (ABS) Neutrophils | 0
  CBC: ABS Lymphocytes | 0
  CBC: ABS Monocytes | 0
  CBC: Neutrophils | 0
  CBC: Lymphocytes | 0
  CMP: Serum Creatinine | 0
  CMP: Creatinine Clearance | 0
  CMP: ALT (SGPT) | 3
  CMP: AST (SGOT) | 2
  CMP: Total Bilirubin | 0
  CMP: Direct Bilirubin | 0
  CMP: Blood Urea Nitrogen (BUN) | 0
  CMP: Albumin | 0
  CMP: Alkaline Phosphate | 2
  CMP: Glucose | 0
  CMP: Calcium | 0
  CMP: Carbon Dioxide | 0
  CMP: Chloride | 0
  CMP: Potassium | 0
  CMP: Sodium | 1
  UA: Specific Gravity | 0
  UA: PH | 0
  UA: Leukocyte Esterase | 42
  UA: Nitrite | 6
  UA: Protein | 32
  UA: Glucose | 5
  UA: Ketones | 19
  UA: Urobilinogen | 1
  UA: Bilirubin | 1
  UA: Blood | 22
  AED: Phenobarbital Level | 0
  AED: Primidone Level | 0
  AED: Klonopin Level | 0
  AED: Clobazam Level | 0
  AED: Desmethylclobazam Level | 0
  AED: Lorazepam Level | 0
  AED: Phenytoin Level | 0
  AED: Carbamazepine Level | 0
  AED: Clorazepate Level | 0
  AED: Valproate Level | 0
  AED: Felbamate Level | 0
  AED: Gabapentin Level | 0
  AED: Lamotrigine Level | 0
  AED: Levetiracetam Level | 0
  AED: Oxcarbazepine Level | 0
  AED: Ethosuximide Level | 0
  AED: Tiagabine Level | 0
  AED: Topiramate Level | 0
  AED: Vigabatrin Level | 0
  AED: Zonisamide Level | 0
  AED: Eslicarbazepine Level | 0
  AED: Ezogabine Level | 0
  AED: Pregabalin Level | 0
  AED: Perampanel Level | 0
  AED: Rufinamide Level | 0
  AED: Brivaracetam Level | 0
  AED: Lacosamide Level | 0
  AED: Diazepam Level | 0

4. Secondary Outcome: Change in Seizure Frequency as Measured in Total Number of Seizures Per Month.
Description: Participants were given seizure diary logs and dairy data collection was done at study clinic visits. Data was recorded and stored in the UAB RedCap System. The analysis plan was to assess the pattern of change in seizure frequency over time, relative to baseline, following CBD exposure. Since the baseline measure was reported at the time of screening, there was some tendency to overestimate the frequency of seizures in the historically reported interval. This was examined by comparing the initial study visits improvement versus the pattern of control over time, and was assessed using graphic techniques and summary statistics.
Time Frame: For 1 Year following Enrollment
Population: Per protocol, after all participants have been enrolled and followed for 1 year. Number of participants analyzed differed because: 1) Those who responded to a certain CBD dose had fewer monthly visits; 2) Those who decided to continue on the same CBD dose had fewer monthly visits; or 3) Withdrawal prior to 1 year following enrollment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: number of seizures/month
Arm/Group | Epidiolex
Number analyzed (Participants) | 80
number of seizures/month
  Month 1 vs Baseline: number analyzed (Participants) | 79
  Month 1 vs Baseline | 0.73 [0.68 to 0.79]
  Month 2 vs Baseline: number analyzed (Participants) | 78
  Month 2 vs Baseline | 0.56 [0.49 to 0.64]
  Month 3 vs Baseline: number analyzed (Participants) | 77
  Month 3 vs Baseline | 0.47 [0.4 to 0.55]
  Month 4 vs Baseline: number analyzed (Participants) | 68
  Month 4 vs Baseline | 0.44 [0.37 to 0.52]
  Month 5 vs Baseline: number analyzed (Participants) | 51
  Month 5 vs Baseline | 0.44 [0.38 to 0.52]
  Month 6 vs Baseline: number analyzed (Participants) | 57
  Month 6 vs Baseline | 0.47 [0.4 to 0.54]
  Month 7 vs Baseline: number analyzed (Participants) | 46
  Month 7 vs Baseline | 0.48 [0.41 to 0.56]
  Month 8 vs Baseline: number analyzed (Participants) | 39
  Month 8 vs Baseline | 0.49 [0.42 to 0.56]
  Month 9 vs Baseline: number analyzed (Participants) | 41
  Month 9 vs Baseline | 0.49 [0.42 to 0.56]
  Month 10 vs Baseline: number analyzed (Participants) | 35
  Month 10 vs Baseline | 0.48 [0.41 to 0.56]
  Month 11 vs Baseline: number analyzed (Participants) | 35
  Month 11 vs Baseline | 0.48 [0.4 to 0.57]
  Month 12 vs Baseline: number analyzed (Participants) | 34
  Month 12 vs Baseline | 0.47 [0.38 to 0.58]
Statistical Analysis 1: Comparison: Epidiolex; Null hypothesis is that there was no change in seizure frequency between any two assessment time points during this period of analysis. Alternative hypothesis is that there were two or more assessment time points for which change in seizure frequency was different from zero; Test type: Other — Single group; p < 0.0001, Wilcoxon (Mann-Whitney) — P-value reported above is the global test for change in seizure frequency over a 12-month period; Wilcoxon signed rank test with Bonferonni multiple comparison correction was used as a post-hoc analysis to indicate direction of change; Generalized least squares statistical techniques were used for modeling longitudinal data after normality of seizure frequency outcome measures were achieved through log-transformations methods. The following baseline clinical variables were adjusted for: AEDs, AEDs tried, epileptic surgery, and gender. Reported results were geometric least squares mean and its associated 95% Confidence Interval. Percentage reduction in seizure frequency relative to baseline were obtained by subtracting from 1 and then multiplying by 100 at all post-baseline timepoints

5. Secondary Outcome: Change in Seizure Severity Measured by the Chalfont Seizure Severity Scale (Duncan & Sander, 1991, JNNP).
Description: Seizure severity was collected during study clinic and phone visits using the Chalfont Seizure Severity Scale (CSSS) (Duncan & Sander, 1991, JNNP) through verbal reporting. The CSSS measured components of seizures most disturbing or disruptive to the participants. The total scores for a given seizure type was its severity score. High scores indicated high severity of the seizures (no fixed maximum value), while a score of zero indicated low severity. Scores were recorded and stored in the UAB RedCap System. The analysis plan was to assess the pattern of change in seizure severity scores over time, relative to baseline, following CBD exposure. Since the baseline measure was reported at the time of screening, there was some tendency to overestimate the severity of seizures in the historically reported interval. This was examined by comparing the initial study visits improvement versus the pattern of control over time, and was assessed using graphic techniques and summary statistics.
Time Frame: For 1 Year following Enrollment
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Epidiolex
Number analyzed (Participants) | 80
scores on a scale
  Month 1 vs Baseline: number analyzed (Participants) | 79
  Month 1 vs Baseline | 0.53 [0.47 to 0.61]
  Month 2 vs Baseline: number analyzed (Participants) | 78
  Month 2 vs Baseline | 0.32 [0.25 to 0.4]
  Month 3 vs Baseline: number analyzed (Participants) | 77
  Month 3 vs Baseline | 0.23 [0.17 to 0.31]
  Month 4 vs Baseline: number analyzed (Participants) | 68
  Month 4 vs Baseline | 0.22 [0.16 to 0.29]
  Month 5 vs Baseline: number analyzed (Participants) | 51
  Month 5 vs Baseline | 0.24 [0.18 to 0.32]
  Month 6 vs Baseline: number analyzed (Participants) | 57
  Month 6 vs Baseline | 0.28 [0.21 to 0.36]
  Month 7 vs Baseline: number analyzed (Participants) | 46
  Month 7 vs Baseline | 0.29 [0.22 to 0.38]
  Month 8 vs Baseline: number analyzed (Participants) | 39
  Month 8 vs Baseline | 0.28 [0.22 to 0.36]
  Month 9 vs Baseline: number analyzed (Participants) | 41
  Month 9 vs Baseline | 0.25 [0.2 to 0.33]
  Month 10 vs Baseline: number analyzed (Participants) | 35
  Month 10 vs Baseline | 0.22 [0.17 to 0.29]
  Month 11 vs Baseline: number analyzed (Participants) | 35
  Month 11 vs Baseline | 0.19 [0.14 to 0.25]
  Month 12 vs Baseline: number analyzed (Participants) | 34
  Month 12 vs Baseline | 0.16 [0.11 to 0.23]
Statistical Analysis 1: Comparison: Epidiolex; Null hypothesis is that there was no change in seizure severity scores between any two assessment time points during this period of analysis. Alternative hypothesis is that there were two or more assessment time points for which change in seizure severity scores was different from zero; Test type: Other — Single group; p < 0.0001, Wilcoxon (Mann-Whitney) — P-value reported above is the global test for change in seizure severity scores over a 12-month period; [statistical method as in outcome 4, analysis 1]; Generalized least squares statistical techniques were used for modeling longitudinal data after normality of seizure severity score outcome measures were achieved through log-transformations methods. The following baseline clinical variables were adjusted for: AEDs, AEDs tried, epileptic surgery, and gender. Reported results were geometric least squares mean and its associated 95% Confidence Interval. Percentage reduction in seizure severity relative to baseline were obtained by subtracting from 1 and then multiplying by 100 at all post-baseline timepoints

ADVERSE EVENTS:
Time Frame: For 1 Year following Enrollment
Description: Adverse events and severe adverse events were collected and reported in all enrolled participants who received study drug. The Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03 was used to determine clinical significance. Adverse events categorized as a grade 3 or above was considered clinically significant. Adverse events grade 4 or above was considered severe adverse events.
Arm/Group | Epidiolex
All-Cause Mortality (participants affected / at risk) | 1/80
Serious Adverse Events (participants affected / at risk) | 14/80
Other Adverse Events (participants affected / at risk) | 73/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidiolex (N=80)
Abnormal liver function panel (Blood and lymphatic system disorders) | 2 (8) — Elevated ALT, Elevated AST
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Esophageal spasm (Gastrointestinal disorders) | 1 (1)
Hospital admission (General disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
Vomiting (Hepatobiliary disorders) | 1 (1)
Nausea (Hepatobiliary disorders) | 1 (1)
Fracture (seizure-related) (Injury, poisoning and procedural complications) | 3 (14)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Status epilepticus (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (5)
Diarrhea (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidiolex (N=80)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (2)
Abnormal liver function panel (Blood and lymphatic system disorders) | 4 (13)
Leukopenia (Blood and lymphatic system disorders) | 1 (18)
Hyponatremia (Blood and lymphatic system disorders) | 4 (12)
Increased International Normalized Ratio (INR) (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Conjuntivitis (Eye disorders) | 1 (2)
Allergic conjunctivitis (Eye disorders) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 53 (428)
Constipation (Gastrointestinal disorders) | 2 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (5)
Belching (Gastrointestinal disorders) | 1 (5)
Hemorrhoid fissure (Gastrointestinal disorders) | 1 (1)
Emergency room visit (General disorders) | 1 (1)
Weight loss (General disorders) | 14 (51)
Weight gain (General disorders) | 2 (16)
Hair loss (General disorders) | 7 (34)
Investigational product complaint (General disorders) | 1 (1) — Reported study drug tasted like cigarettes
Arachnidism (General disorders) | 1 (1)
Friction burn (General disorders) | 1 (1)
Cyst (General disorders) | 2 (4)
Anorexia (Hepatobiliary disorders) | 1 (13)
Decreased appetite (Hepatobiliary disorders) | 10 (49)
Abdominal pain (Hepatobiliary disorders) | 4 (24)
Nausea (Hepatobiliary disorders) | 7 (14)
Mycoplasma (Infections and infestations) | 1 (1)
Flu (Infections and infestations) | 2 (3)
Viral gastroenteritis (Infections and infestations) | 2 (2)
Common cold (Infections and infestations) | 10 (18)
Ear infection (Infections and infestations) | 3 (6)
Fever (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Strep throat (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 5 (10)
Staph infection of the skin (Infections and infestations) | 1 (2)
Fracture (seizure-related) (Injury, poisoning and procedural complications) | 1 (9)
B-12 deficiency (Metabolism and nutrition disorders) | 1 (7)
Lower body pain (Musculoskeletal and connective tissue disorders) | 3 (9) — Includes leg, knee, lower back
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Sedation (Nervous system disorders) | 15 (73)
Insomnia (Nervous system disorders) | 4 (12)
Dizziness (Nervous system disorders) | 9 (22)
Eyes rolling back (Nervous system disorders) | 1 (3) — Seizure-related
Sleep disturbance (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 2 (3)
Double vision (Nervous system disorders) | 3 (3)
Lethargic (Nervous system disorders) | 6 (27)
Hand tremors (Nervous system disorders) | 1 (2)
Fall (seizure-related) (Nervous system disorders) | 4 (6)
Fall (unrelated to seizure) (Nervous system disorders) | 1 (1)
Increased seizure frequency (Nervous system disorders) | 2 (2)
Depression/mood issues (Psychiatric disorders) | 6 (27)
Kidney stones (Renal and urinary disorders) | 1 (3)
Urinary tract infection (Renal and urinary disorders) | 5 (8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 1 (12)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (4)
Worsening uticaria (Skin and subcutaneous tissue disorders) | 1 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (10)
Ingrown toenail (Skin and subcutaneous tissue disorders) | 1 (2)
Buttock contusion (Skin and subcutaneous tissue disorders) | 1 (2)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (4)
Gallbladder removal (Surgical and medical procedures) | 1 (1)
Headaches (Vascular disorders) | 9 (31)
Gastroenteritis (Infections and infestations) | 2 (3)
Lacerations (Skin and subcutaneous tissue disorders) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Flexible dosing schedule; Over- or underreporting of seizure frequency and severity that may reflect patients' or caregivers' desires to qualify or remain in the study; Non-normality of the data; Early withdrawal of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02700412/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT02700412/SAP_001.pdf